CLINICAL TRIAL: NCT03681171
Title: A Pilot Study of a Therapeutic Dance Intervention for Children With Cerebral Palsy
Brief Title: Therapeutic Dance Intervention for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shlomit Aizik (Other)
Responsible Party: Sponsor-Investigator, Shlomit Aizik, Associate Professor, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-2682
Record Dates: First submitted 2018-08-30; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with CP (Experimental): Children with CP (9-15 years old) participated in a therapeutic dance program to improve physical, physiological and cognitive outcomes.
  Interventions: Other: Therapeutic Dance

INTERVENTIONS:
Other: Therapeutic Dance — Participants attended therapeutic ballet sessions three times per week for six weeks.

SUMMARY:
Children with cerebral palsy (CP) have motor impairments that make it challenging for them to participate in standard physical activity (PA) programs. There is a need to evaluate adapted PA programs for this population. Dance can promote coordination, posture, muscle strength, motor learning, and executive functioning. This pilot study evaluated the feasibility and the effects of a new therapeutic ballet intervention specifically designed for children with CP on physiological and executive functions outcomes.

DETAILED DESCRIPTION:
8 children with CP (9-14y/o; 75% female) participated in a six-week therapeutic ballet program. Participants had body composition (DXA), muscle strength (hand-grip dynamometer), habitual physical activity, gait and selective motor control functions, and executive function tasks before and after the intervention. Follow-up assessments of habitual physical activity, gait and executive functions were completed four to five week post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy spastic diplegia and/or hemiplegia
* Absence of health problems that would preclude participation in exercise
* Male or female age 9 - 15 years inclusive at the time of consent
* Minimum level of intellectual functioning (e.g., as determined by an IQ score of 80 or above or other education placement and testing indicating sufficient understanding)
* Ability to complete study measures at the assessment
* Ability to participate in dance classes conducted in English
* Interest in learning ballet
* Intact vision
* Intact hearing
* Able to ambulate independently in the community with or without a device
* Intact proprioception in lower extremities
* Able to complete assessment measures and consents in English
* Referral from the child's pediatrician or other physician indicating that the child is physically able to participate in an exercise intervention

Exclusion Criteria:

* Children with a current diagnosis of severe Major Depressive Disorder
* Generalized Anxiety Disorder
* Epilepsy
* Autism
* Other major medical conditions that prohibit full participation and children with severe developmental disorders (e.g., mental retardation, severe autism) or with physical impairments that prohibit full participation were excluded from the study.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2016-06-25 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Gait (GAITRite© system) | 12 weeks
  Assessment before an immediately after six-week therapeutic ballet program and 4-5 weeks post intervention
Executive Functions measured by Hearts and Flowers Flanker Tasks | 12 weeks
  Measures attention and working memory before an immediately after six-week therapeutic ballet program and 4-5 weeks post intervention.
Executive Functions measured by Stroop Colored Word Test | 12 weeks
  Measures inhibitory control before an immediately after six-week therapeutic ballet program and 4-5 weeks post intervention.
Executive Functions measured by BRIEF (Parent Questionnaire) | 12 weeks
  An 86-item questionnaire

SECONDARY OUTCOMES:
Body Composition Dual X-ray Absorptiometry, DXA scan before and after six-week therapeutic ballet program. | 8 weeks
  Assessment of Lean Body Mass
Body Composition Dual X-ray Absorptiometry, DXA scan before and after six-week therapeutic ballet program. | 8 weeks
  Assessment of Percent Body Fat
Body Composition Dual X-ray Absorptiometry, DXA scan before and after six-week therapeutic ballet program. | 8 weeks
  Assessment of bone density
Muscle Strength | 8 weeks
  Handgrip (evaluated maximum isometric strength (Kg) before and after six-week therapeutic ballet program.
CBC | 8 weeks
  Includes hemoglobin measures for anemia and inflammation factors
Lipid Panel | 8 weeks
  CVD risk factors (lipid screen ) before and after six-week therapeutic ballet program
Habitual Physical Activity assessment | 12 weeks
  Physical activity was measured using ActiGraph accelerometers before and immediately after six-week therapeutic ballet program and 4-5 weeks post intervention.
Social and Emotional Functioning measured by Self-Efficacy Survey (Child) | 8 weeks
  Measures individual perceptions of one's capacity to manage one's functioning and control over events before and after six-week therapeutic ballet program.
Social and Emotional Functioning measured by Self-Perception Profile for Children | 8 weeks
  Measures Scholastic Competence, Athletic Competence, Social Competence, Physical Appearance, and Behavioral Conduct.
Social and Emotional Functioning measured by Positive Affect Survey. | 8 weeks
  Measures feelings of pleasurable engagement with the environment (happiness, joy, excitement, engagement).
Social and Emotional Functioning measured by Perceived Stress Self-Report Scale | 8 weeks
  Asks participants to rate how they have felt over the last month
Social and Emotional Functioning measured by Strengths and Difficulties Questionnaire (SDQ) | 8 weeks
  SDQ is a brief questionnaire that assesses children's emotional problems

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Aizik, PhD, Study Director — University of California, Irvine

REFERENCES:
- [Derived] Lakes KD, Sharp K, Grant-Beuttler M, Neville R, Haddad F, Sunico R, Ho D, Schneider M, Sawitz S, Paulsen J, Caputo K, Lu KD, Aminian A, Lopez-Ortiz C, Radom-Aizik S. A Six Week Therapeutic Ballet Intervention Improved Gait and Inhibitory Control in Children With Cerebral Palsy-A Pilot Study. Front Public Health. 2019 Jun 25;7:137. doi: 10.3389/fpubh.2019.00137. eCollection 2019. PMID 31294009